CLINICAL TRIAL: NCT01747395
Title: Effects of Aerobic Exercise Training Associated With Inspiratory Muscle Training in Patients With Heart Failure
Brief Title: Exercise Training Associated With Inspiratory Muscle Training in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Patricia Fernandes Trevizan, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICRESP814/10
Record Dates: First submitted 2012-12-06; First posted 2012-12-11 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Exercise and Physical Fitness
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Group (No Intervention): No exercise group (sedentary)
- Aerobic Exercise Training (Experimental): Group undergoing isolate aerobic exercise training 3 times/week, during 40 minutes, for 04 mouths
  Interventions: Other: Exercise training
- Inspiratory Muscle Training (Experimental): Group undergoing isolate inspiratory muscle training 7 times/week, during 30 minutes, for 04 mouths
  Interventions: Other: Exercise training
- Aerobic+Inspiratory Muscle Training (Experimental): Group undergoing aerobic exercise training (3 times/week during 40 minutes) associate inspiratory muscle training (7 times/week during 30 minutes) for 04 mounths
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — The heart failure patients are subjected to differents protocols of physical training
  Arms: Aerobic Exercise Training; Aerobic+Inspiratory Muscle Training; Inspiratory Muscle Training

SUMMARY:
The investigators hypothesize that aerobic exercise training associated with respiratory muscle training will cause additional benefits compared to isolated exercise training or respiratory training in chronic heart failure patients.

DETAILED DESCRIPTION:
The investigators hypothesize that aerobic exercise training associated with respiratory muscle training will cause additional benefits in the autonomic control and respiratory function compared to isolated exercise training or respiratory training in chronic heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systolic heart failure and New York Heart Association (NYHA) class II-III
* Left ventricular ejection fraction less than 40%
* Peak Oxygen Consumption less than 20 ml/Kg/min

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease
* Neuromuscular, Orthopedic, Neurologic and Neoplastic Diseases
* Recent myocardial infarction or cardiac surgery (less than 6 months)
* Unstable angina pectoris
* Atrial Fibrillation
* Pacemakers users
* Actual Smoker
* Pregnant
* Changing medication or hospital admission

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2020-04 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Autonomic control | 4 months
  Exercise training associated with inspiratory muscle training will reduce sympathetic nerve activity.

SECONDARY OUTCOMES:
Functional Capacity | 4 months
  Exercise training associated with inspiratory muscle training will improve peak oxygen consumption
Quality of life | 4 months
  Exercise training associated with inspiratory muscle training will improve quality of life
Blood inflammatory markers | 4 months
  Exercise training associated with inspiratory muscle training will reduces blood inflammatory markers
Muscular evaluation | 4 months
  Exercise training associated with inspiratory muscle training will increase skeletal muscle strength
Respiratoy muscle function | 4 months
  Exercise training associated with inspiratory muscle training will increase inspitarory muscle strength and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Eduardo Negrão, Principal Investigator — InCor, HCFMUSP
Locations (1):
- Instituto do Coração - HC/FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antunes-Correa LM, Trevizan PF, Bacurau AVN, Ferreira-Santos L, Gomes JLP, Urias U, Oliveira PA, Alves MJNN, de Almeida DR, Brum PC, Oliveira EM, Hajjar L, Kalil Filho R, Negrao CE. Effects of aerobic and inspiratory training on skeletal muscle microRNA-1 and downstream-associated pathways in patients with heart failure. J Cachexia Sarcopenia Muscle. 2020 Feb;11(1):89-102. doi: 10.1002/jcsm.12495. Epub 2019 Nov 19. PMID 31743617